CLINICAL TRIAL: NCT05836688
Title: A Biobehavioral Intervention to Reduce Adverse Outcomes in Young Adult Testicular Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Michael Hoyt, Associate Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20205812; 1R01CA276143-01A1 (NIH)
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Testicular Cancer
MeSH Terms: conditions — Testicular Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Goal-Focused Emotion-Regulation Therapy (GET) (Experimental): A novel behavioral intervention to enhance self-regulation through improved goal navigation skills, improved sense of purpose, and better ability to regulate emotional responses in young adults with testicular cancer.
  Interventions: Behavioral: Goal-Focused Emotion-Regulation Therapy (GET)
- Individual Supportive Listening (Active Comparator): Supportive therapy will be non-directive and will primarily reinforce a patient's ability to manage stressors through attentively listening and encouraging expression of thoughts and feelings, assisting the individual to gain a greater understanding of their situation and alternatives, and helping to buttress the individual's self-esteem and resilience.
  Interventions: Behavioral: Individual Supportive Listening

INTERVENTIONS:
Behavioral: Goal-Focused Emotion-Regulation Therapy (GET) — Patients will be asked to identify value-derived goals (i.e., goals for the most important domains of one's life) and ones sufficiently important to sustain movement toward them in the short-term future. Patients will discuss their goal possibilities, providing a forum to ensure that goals are manageable and consistent with identified values. Patients will learn strategies to refine their goals (e.g., approaching goals rather than avoiding obstacles, defining markers of progress), generate pathways to goals, and address potential obstacles and blockages. The overall goal is to enhance self-regulation through improved goal navigation skills, improved sense of meaning and purpose, and better ability to regulate specific emotional responses.
  Arms: Goal-Focused Emotion-Regulation Therapy (GET)
Behavioral: Individual Supportive Listening — ISL sessions will be matched in terms of time and attention. Supportive therapy will be non-directive and will primarily reinforce a patient's ability to manage stressors through attentively listening and encouraging expression of thoughts and feelings, assisting the individual to gain a greater understanding of their situation and alternatives, and helping to buttress the individual's self-esteem and resilience. This will be delivered in the same manner as GET (individually) and is a common, non-directive control method in intervention research.
  Arms: Individual Supportive Listening

SUMMARY:
This study is a randomized controlled biobehavioral efficacy trial designed to investigate the feasibility and acceptability of a novel intervention, Goal-focused Emotion-Regulation Therapy (GET) aimed at improving distress symptoms, emotion regulation, goal navigation skills, and stress-sensitive biomarkers in young adult testicular cancer patients.

Participants will be randomized to receive six sessions of GET or Individual Supportive Listening (ISL) delivered over eight weeks. In addition to indicators of intervention feasibility, the investigators will measure primary (depressive and anxiety symptoms) and secondary (emotion regulation and goal navigation skills, career confusion) psychological outcomes prior to (T0), immediately after (T1), twelve weeks after intervention (T2) and 24 weeks after the intervention (T3). Additionally, identified biomarkers will be measured at baseline and at T1, T2, and T3.

DETAILED DESCRIPTION:
Testicular cancer diagnosis and treatment, especially given its threat to sexuality and reproductive health, can be distressing in the formative period of young adulthood. Cohort studies reveal the prevalence of depressive symptoms in testicular cancer exceeds the general population. In fact, the majority of young adult cancer survivors will experience impairing, distressing, and modifiable physical, behavioral, and psychosocial adverse outcomes that persist long after the completion of primary medical treatment. These include psychological distress, impairment in the navigation and pursuit of life goals, persistent side effects, elevated risk of secondary malignancies and chronic illness, and biobehavioral burden (e.g., enhanced inflammation, dysregulated stress hormones) which influence morbidity and disease-related vulnerabilities. However, few targeted, effective interventions exist to assist young survivors in re-negotiating life goals and regulating cancer-related emotions and none focus on reducing the burden of morbidity via biobehavioral mechanisms.

Young or "emerging" adulthood is a period marked by goal attainment. Chronic illness experienced as "off time" in the lifespan interrupts goal pursuits and threatens valued life directions. As young adults return to goal pursuits, re-entry to post-cancer life can be a critical point in the survivorship trajectory. Behavioral intervention at this time is well positioned to confer longer-term impact. Emergent from our group's preliminary research, we developed and pilot-tested Goal-focused Emotion-Regulation Therapy (GET) as a novel behavioral intervention to enhance self-regulation through improved goal navigation skills, improved sense of purpose, and better ability to regulate emotional responses in young adults with testicular cancer. GET is a promising candidate intervention to address the mechanisms likely complicating the resolution of cancer-related burden.

Responsive the need for feasible, effective, and scalable interventions, we will randomly allocate 250 young adult (ages 18 -39) testicular cancer patients to 6 sessions of GET or ISL, and evaluate primary and secondary outcomes at baseline, post-treatment, 3-month follow-up, and 6-months follow-up. We predict that GET will be associated with superior distress outcomes and comparatively greater reductions in adverse biobehavioral indicators (dysregulated diurnal stress hormones, elevated systemic inflammation), and these advantages will be maintained at three- and six-months following intervention. The intervention will be delivered via an interactive video platform to enhance access. An additional exploratory aim focuses on potential epigenetic vulnerabilities, to understand how environmental influences (via DNA methylation) on genes implicated in stress reactivity and mood regulation are related to cancer adjustment and intervention response.

This study capitalizes on the study team's unique expertise in biobehavioral oncology and salivary bioscience to test a novel behavioral intervention for young adult survivors. It has potential to understand how to alter proximal behavioral, biological, and psychological factors that underscore long term adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 39 years at time of consent
* A confirmed diagnosis of testis cancer (any stage)
* Completion of chemotherapy for testis cancer within 4 years prior to consent
* A score of >4 on the Distress Thermometer
* English fluency, as per medical record documenting preferred language or in the judgment of the investigator
* Spanish fluency, as per medical record documenting preferred language or in the judgment of the investigator
* Able to perform informed consent

Exclusion Criteria:

* Lifetime history of psychiatric of cognitive disturbance as per self-report or medical record
* In the judgment of the consenting professional, is unable to provide informed consent and complete study sessions and assessment
* As per self-report, has medical conditions that affect the immune system and would confound immune evaluation (e.g., autoimmune disorder, inflammatory disease; uncontrolled thyroid disease; active infection; myocardial infarction or stroke in the last 6 months; Type I diabetes; acute hepatitis; recent vaccination for viral disease)
* Regular smoker (daily use)

Ages: 18 Years to 39 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Change in Hospital Anxiety and Depression Scale (HADS) | Change from Baseline (T0) to intervention completion (~8 weeks), to 3-month post-intervention (~20 weeks), and to 6-month post-intervention (~32 weeks)
  The HADS was developed to assess anxiety and depression in medical patients. It purposefully excluded somatic symptoms (e.g., sleep disturbance) to reduce confounding psychological symptoms with disease or treatment. The HADS has become a "benchmark" measure of anxiety and depression among diverse clinical and nonclinical hospital populations, including individuals diagnosed with cancer. The HADS is a 14-item self-administered questionnaire, with 7 items assigned to each the HADS-Anxiety and HADS-Depression subscales. Each item is rated on a 4-point response scale (from 0 to 3). Subscale scores are typically categorized to indicate the level of anxiety or depression experienced where scores of less than 8 are categorized as normal, scores of 8-10 as borderline, and scores of 11-21 as clinical. A number of psychometric studies have established the scale's strengths, including its brevity, reliability, and validity and availability of comparison scores across different populations.
Change in Systemic Pro-inflammatory Cytokine Levels (IL-6, IL-1ra, C-reactive Protein [CRP], sTNFαRII) | Change from Baseline (T0) to intervention completion (~8 weeks), to 3-month post-intervention (~20 weeks), and to 6-month post-intervention (~32 weeks)
  The investigators will focus on four biomarkers, IL-6, IL-1ra, CRP, sTNFαRII, that indicate systemic inflammation and are associated with distress symptoms and emotion regulation. Levels will be assessed from plasma. Cytokine levels will be determined by immunosorbent assay (ELISA) according to assay manufacturer's protocols. All samples will be run in duplicate, and assays will be repeated on two separate days; intra-assay and interassay mean levels will be used in all analyses.
Change in Salivary Diurnal Cortisol Slope and Daily Output | Change from Baseline (T0) to intervention completion (~8 weeks), to 3-month post-intervention (~20 weeks), and to 6-month post-intervention (~32 weeks)
  Diurnal rhythm in salivary cortisol will be measured over three days at each assessment. Participants will collect saliva samples in their natural environment upon awakening, 30 minutes later, 8 hours later, and at bedtime. Participants will complete a diary to assess relevant health behaviors (e.g., caffeine, tobacco, alcohol consumption; physical activity, sleep) as well as daily stress. They will be instructed to avoid brushing their teeth, eating, or drinking within 20 minutes before sampling. Participants will keep samples refrigerated prior to returning them to the research laboratory and returned salivettes will be stored in a -20-degree Celsius freezer until analyzed. Salivary cortisol will be analyzed with a time-resolved fluorescence immunoassay. Several indices will be computed including diurnal slope, area under the daily curve, cortisol awakening response, and total daily cortisol output.

SECONDARY OUTCOMES:
Change in Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being (FACIT-Sp) Subscale Score | Change from Baseline (T0) to intervention completion (~8 weeks), to 3-month post-intervention (~20 weeks), and to 6-month post-intervention (~32 weeks)
  A 12-item questionnaire that measures spiritual well-being in people with cancer and other chronic illnesses. The FACIT-Sp-12 is part of the larger Functional Assessment of Chronic Illness Therapy (FACIT) measurement system that assesses multidimensional HRQOL. It asks patients to describe aspects of spirituality and/or religious faith that contribute to HRQOL over the past 7 days. The measure was originally developed with 2 components or factors of a total (overall) score: a 4-item Faith component (e.g. I find comfort in my faith or spiritual beliefs), and an 8-item Meaning/Peace component (e.g. I feel a sense of purpose in my life, I feel peaceful).
Change in Career Thoughts Inventory (CTI) Global Score | Change from Baseline (T0) to intervention completion (~8 weeks), to 3-month post-intervention (~20 weeks), and to 6-month post-intervention (~32 weeks)
  The CTI (Sampson et al., 1996) is a 48-item self-administered instrument that measures an individual's level of dysfunctional thinking in career decision-making and career problem-solving. The CTI is normed on adults and broadly used in the context of I/O Psychology. Items are rated on a 4-point Likert scale ranging from 0 (strongly disagree) to 3 (strongly agree). CTI total score provides information about an individual's overall level of dysfunctional career thoughts, However, the CTI has three subscales: Decision-Making Confusion (difficulties with initiating or sustaining a career choice), Commitment Anxiety (difficulties with making a commitment to a career choice), and External Conflict (difficulties with balancing one's ideas with the ideas from others). The CTI has sound evidence for its content, construct, and criterion-related validity (Peila-Shuster & Feller, 2013; Sampson et al., 1996).
Change in Emotion Regulation Questionnaire (ERQ) Scale Scores | Change from Baseline (T0) to intervention completion (~8 weeks), to 3-month post-intervention (~20 weeks), and to 6-month post-intervention (~32 weeks)
  Emotion regulation skills will be measured by the Emotion Regulation Questionnaire (ERQ). The ERQ is a widely used 10-item scale designed to measure respondents' tendency to regulate their emotions in two ways: (1) Cognitive Reappraisal and (2) Expressive Suppression. Respondents answer each item on a 7-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree). The ERQ is widely used in the context of clinical treatment trials and has well established validity, reliability, and factor structure (Goldin, Manber-Ball, Werner, Heimberg, & Gross, 2009; Gross & John, 2003).
Change in Cancer Assessment for Young Adults (CAYA-T) - Goal Navigation Score | Change from Baseline (T0) to intervention completion (~8 weeks), to 3-month post-intervention (~20 weeks), and to 6-month post-intervention (~32 weeks)
  Goal navigation capacity includes elements of goal setting, goal clarification, goal adjustment, and goal initiation. It will be measured by the Goal Navigation subscale of the Cancer Assessment for Young Adults -Testicular (CAYA-T) (Hoyt et al., 2013). The scale is composed of five items (e.g., "I am able to identify goals in my life", "I know what steps to take to make progress toward my goals", and "I am able to redirect my energy when I feel my life isn't going in the right direction"). Participants indicate how often each item is true of them over the past 7 days on a 3-point response scale ranging from 0 (None of the time) to 2 (Much or most of the time). Criterion, construct, and procedural validity have been established with young adult testicular cancer survivors.
Change in Emotional Approach Coping Questionnaire (EAC) Scale Scores | Change from Baseline (T0) to intervention completion (~8 weeks), to 3-month post-intervention (~20 weeks), and to 6-month post-intervention (~32 weeks)
  The EAC Scale is an 8-question, patient-rated, self-report scale designed to measure emotional coping. Participants are asked to rate their usual response to stress by rating each item on a 4-point Likert scale (1 = "I usually don't do this at all" to 4 = "I usually do this a lot"). The scores for the EAC range from 0 to 32, with lower scores representing poorer emotional coping.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Hoyt, PhD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hoyt MA, Wang AW, Ryan SJ, Breen EC, Cheavens JS, Nelson CJ. Goal-Focused Emotion-Regulation Therapy (GET) for young adult survivors of testicular cancer: a pilot randomized controlled trial of a biobehavioral intervention protocol. Trials. 2020 Apr 14;21(1):325. doi: 10.1186/s13063-020-04242-0. PMID 32290859
- [Background] Hoyt MA, Nelson CJ. Goal-focused Emotion-Regulation Therapy for young adult survivors of testicular cancer: Feasibility of a behavioral intervention. Contemp Clin Trials Commun. 2020 Aug 21;19:100648. doi: 10.1016/j.conctc.2020.100648. eCollection 2020 Sep. PMID 32913918
- [Background] Hoyt MA, Wang AW, Breen EC, Nelson CJ. A Randomized Controlled Trial of Goal-Focused Emotion-Regulation Therapy for Young Adult Survivors of Testicular Cancer: Effects on Salivary and Inflammatory Stress Markers. Am J Mens Health. 2021 Sep-Oct;15(5):15579883211044557. doi: 10.1177/15579883211044557. PMID 34514890